CLINICAL TRIAL: NCT07181161
Title: A Modular Phase I/IIa, Open-label, Multi-centre Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of AZD0516 as Monotherapy and in Combination With Anti-cancer Agents in Participants With Metastatic Prostate Cancer
Brief Title: Study of AZD0516 as Monotherapy and in Combination in Participants With Metastatic Prostate Cancer
Acronym: SEACLIFF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9520C00001; 2024-520026-11-00 (Other: EU CT Number)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer; Dose escalation study; Anti-cancer agents; Antibody-drug conjugate; Anti-Six-transmembrane epithelial antigen of the prostate 2 (anti-STEAP2); Metastatic castration resistant prostate cancer (mCRPC); AZD0516
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: AZD0516 monotherapy (Experimental): Participants with mCRPC will receive AZD0516 monotherapy.
  Interventions: Drug: AZD0516
- Arm 2: AZD0516 + AZD9574 (Experimental): Participants with mCRPC will receive AZD0516 in combination with AZD9574.
  Interventions: Drug: AZD0516; Drug: AZD9574

INTERVENTIONS:
Drug: AZD0516 — AZD0516 will be administered via intravenous infusion.
Drug: AZD9574 — AZD9574 will be administered orally.
  Arms: Arm 2: AZD0516 + AZD9574

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of AZD0516 as monotherapy and/or in combination with other anti-cancer agents for treatment of metastatic prostate cancer.

DETAILED DESCRIPTION:
This is a first-in-human modular, Phase I/IIa, open-label, multi-centre study of AZD0516 in participants with metastatic prostate cancer. The study will consist of individual modules, each evaluating the safety, tolerability, preliminary efficacy, PK, pharmacodynamic, and immunogenicity of AZD0516.

Module 1: Evaluates AZD0516 as monotherapy. It may include 3 parts, Part A- Dose Escalation, Part B- Dose Optimisation, and Part C- Efficacy Expansion.

Module 2: Evaluates AZD0516 in combination with AZD9574. It may include 2 parts, Part A - Dose Escalation and Part B Dose Optimisation.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic adenocarcinoma of the prostate. Focal high grade neuroendocrine features are permitted.
* Measurable PSA ≥ 1 μg/L (≥ 1 ng/mL).
* Surgically or medically castrated with serum testosterone levels ≤ 50 ng/dL (≤ 1.75 nmol/L) within ≤ 28 days before treatment allocation. Ongoing androgen deprivation therapy (ADT) with a gonadotropin releasing hormone (GnRH) modulator for participants who have not undergone bilateral orchiectomy must be initiated at least 2 weeks prior to consent and must continue throughout the study.
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.
* Adequate organ and marrow function in the absence of blood transfusion or growth factor support (within 21 days prior to the scheduled first dose of study intervention).
* Provision of baseline archival or newly obtained formalin-fixed paraffin-embedded (FFPE) tumour sample is mandatory.
* Documented current evidence of metastatic prostate cancer
* Life expectancy of at least 12 weeks in the opinion of the investigator
* Documented mCRPC progression at screening as assessed by the investigator with at least one of the following criteria:

  1. PSA progression defined by a minimum of 3 rising PSA levels with an interval of ≥ 1 week between each determination. The PSA value at the screening visit should be ≥ 1 μg/L (1 ng/mL).
  2. Radiographic disease progression in soft tissue based on response evaluation criteria in solid tumors (RECIST) v1.1 criteria with or without PSA progression as per prostate cancer working group 3 (PCWG3).
  3. Radiographic disease progression in bone defined as the appearance of 2 or more new bone lesions on a bone scan as per PCWG3 with or without PSA progression.

Main Exclusion Criteria:

* Cancer related spinal cord compression, or brain metastases unless asymptomatic, treated and stable and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent for at least 4 weeks prior to study enrolment.
* History of leptomeningeal carcinomatosis.
* Unresolved toxicities of Grade ≥ 2 (National Cancer Institute Common Terminology Criteria for Adverse Events v5.0) from prior therapy (excluding vitiligo, alopecia, and endocrine disorders that are controlled with replacement hormone therapy).
* Uncontrolled intercurrent illness within the last 12 months.
* Cardiovascular disorder (History of arrhythmia, uncontrolled hypertension, symptomatic hypotension, history of brain perfusion problems, symptomatic heart failure, prior or current cardiomyopathy, severe valvular heart disease)
* History of malignancy
* History of non-infectious interstitial lung disease (ILD)/pneumonitis
* Active infection exclusions, including tuberculosis and infections with Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV).
* Any known predisposition to bleeding
* Clinically severe pulmonary compromise
* Participants with Myelodysplastic syndrome (MDS)/Acute Myeloid Leukemia (AML) or with features suggestive of MDS/AML.
* Previous treatment with a STEAP2 targeting modality, chemotherapeutic agent that inhibits topoisomerase activity or metabolic enzymes.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 177 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-01-18 (Estimated); Study Completion 2029-01-18 (Estimated)

PRIMARY OUTCOMES:
Module 1 and 2: Parts A and B: Number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Event of Special Interests (AESIs) | From Day 1 up to approximately 3 years
  Part A: To assess the safety and tolerability and to determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose for Expansion (RDE) of AZD0516 as monotherapy and in combination with anti-cancer agents.
  Part B: To assess the safety and tolerability of AZD0516 as monotherapy and in combination with anti-cancer agents.
Module 1 and 2: Part A: Number of participants with Dose Limiting Toxicities (DLTs) | From Day 1 up to end of DLT period (approximately 21 days)
  To assess the safety and tolerability of AZD0516 as monotherapy and in combination with anti-cancer agents.
Module 1: Parts B and C and Module 2: Part B: Percentage of participants with Prostate-Specific Antigen (PSA) 50 response rate | Up to approximately 2 years
  The PSA50 response rate is defined as the percentage of participants achieving ≥ 50% decrease in PSA from baseline to the lowest post-baseline PSA result.

SECONDARY OUTCOMES:
Module 1 and 2: Part A: Percentage of participants with PSA50 response rate | Up to approximately 2 years
  The PSA50 response rate is defined as the percentage of participants achieving ≥ 50% decrease in PSA from baseline to the lowest post-baseline PSA result.
Module 1 and 2: Parts A, B and C: Percentage of participants with PSA90 response rate | Up to approximately 2 years
  The PSA90 response rate is defined as the percentage of participants with a confirmed ≥ 90% decrease in PSA from baseline to the lowest post-baseline PSA result.
Module 1 and 2: Parts A, B and C: Time to PSA 50 response (TTPSA50) | Up to approximately 2 years
  The TTPSA response is defined as the time from the date of first dose of study intervention until the date of first documented PSA50 response (≥ 50% decrease in PSA from baseline, respectively) that is confirmed by a second consecutive PSA assessment at least 3 weeks later.
Module 1 and 2: Parts A, B and C: Time to PSA response (TTPSA90) | Up to approximately 2 years
  The TTPSA response is defined as the time from the date of first dose of study intervention until the date of first documented PSA90 response (≥ 90% decrease in PSA from baseline, respectively) that is confirmed by a second consecutive PSA assessment at least 3 weeks later.
Module 1 and 2: Parts A, B and C: Duration of PSA response 50 (DoPSA50) | Up to approximately 2 years
  The DoPSA50 is defined as the time from the date of first documented PSA50 response, that is subsequently confirmed by a second consecutive PSA assessment at least 3 weeks later, until the date of documented PSA progression.
Module 1 and 2: Parts A, B and C: Duration of PSA response 90 (DoPSA90) | Up to approximately 2 years
  The DoPSA90 is defined as the time from the date of first documented PSA90 response, that is subsequently confirmed by a second consecutive PSA assessment at least 3 weeks later, until the date of documented PSA progression.
Module 1 and 2: Parts A, B and C: Percentage of participants with Durable PSA response rate 50 (DRRPSA50) | Up approximately 2 years
  The DRRPSA50 is defined as the percentage of participants who have a documented PSA50 response that is subsequently confirmed by a second consecutive PSA assessment at least 3 weeks later, with a duration of at least 6 months.
Module 1 and 2: Parts A, B and C: Percentage of participants with Durable PSA response rate 90 (DRRPSA90) | Up to approximately 2 years
  The DRRPSA90 is defined as the percentage of participants who have a documented PSA90 response that is subsequently confirmed by a second consecutive PSA assessment at least 3 weeks later, with a duration of at least 6 months.
Module 1 and 2: Parts A, B and C: Time to PSA Progression (TTPSA) | Up to approximately 2 years
  TTPSA progression is defined as time from the date of first dose of study intervention until the date of documented PSA progression or the last PSA result in the absence of progression.
Module 1 and 2: Parts A, B and C: Percentage change from baseline in PSA levels | Up to approximately 2 years
  The percentage change from baseline in PSA levels will be assessed.
Module 1 and 2: Parts A, B and C: Percentage of participants with Overall Response Rate (ORR) | Up to approximately 3 years
  The ORR is defined as the percentage of participants with a confirmed tumour response of Complete Response (CR) or Partial Response (PR).
Module 1 and 2: Parts A, B and C: Percentage of participants with Best Overall Response (BOR) | Up to approximately 3 years
  The BOR is defined as the best overall visit response achieved by participant.
Module 1 and 2: Parts A, B and C: Duration of Response (DoR) | Up to approximately 3 years
  The DoR is defined as the time from the date of first documented objective response (which is subsequently confirmed) until the date of radiographic disease progression or censoring.
Module 1 and 2: Parts A, B and C: Percentage of participants with Durable Response Rate (DRR) | Up to approximately 3 years
  The DRR is defined as the percentage of participants who have a confirmed response with a duration of at least 6 months.
Module 1 and 2: Parts A, B and C: Percentage of participants with Disease Control Rate (DCR) | Up to approximately 3 years
  The DCR is defined as the percentage of participants who have a BOR of confirmed CR or PR or Stable Disease (SD).
Module 1 and 2: Parts A, B and C: Time to Response (TTR) | Up to approximately 3 years
  The TTR is defined as the time from the date of first dose of study intervention until the date of first documented objective response, which is subsequently confirmed.
Module 1 and 2: Parts A, B and C: Percentage Change in Tumour Size | Up to approximately 3 years
  The best percentage change from baseline in tumour size is the largest decrease (or smallest increase) from baseline for a participant, using response evaluation criteria in solid tumors (RECIST) v1.1 assessments.
Module 1 and 2: Parts A, B and C: Radiographic Progression-free Survival (rPFS) | Up to approximately 3 years
  rPFS is defined as the time from date of first dose of study intervention until the date of objective disease progression according to RECIST v1.1 (for soft tissue disease) and prostate cancer working group 3 (PCWG3) criteria (for bone disease) as assessed by the investigator at the local site, or death (by any cause in the absence of progression).
Module 1 and 2: Parts A, B and C: Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from date of first dose of study intervention until death due to any cause.
Module 1 and 2: Part A and B: Changes in Plasma concentration of AZD0516 | From Day 1 up to approximately 3 years
  To characterise the pharmacokinetics (PK) of AZD0516 when given as monotherapy and in combination with anti-cancer agents.
Module 1 and 2: Parts A and B: Area under concentration-time curve (AUC) | From Day 1 up to approximately 3 years
  To characterise the PK (AUC) of AZD0516 when given as monotherapy and in combination with anti-cancer agents.
Module 1 and 2: Parts A and B: Maximum observed drug concentration (Cmax) | From Day 1 up to approximately 3 years
  To characterise the PK (Cmax) of AZD0516 when given as monotherapy and in combination with anti-cancer agents.
Module 1 and 2: Parts A and B: Time to reach maximum observed concentration (tmax) | From Day 1 up to approximately 3 years
  To characterise the PK (tmax) of AZD0516 when given as monotherapy and in combination with anti-cancer agents.
Module 1 and 2: Parts A and B: Tobal Body Clearance (CL) | From Day 1 up to approximately 3 years
  To characterise the PK (CL) of AZD0516 when given as monotherapy and in combination with anti-cancer agents.
Module 1 and 2: Parts A and B: Half-life (t1/2) | From Day 1 up to approximately 3 years
  To characterise the PK (t1/2) of AZD0516 when given as monotherapy and in combination with anti-cancer agents.
Module 1 and 2: Parts A and B: Plasma concentration of total antibody (conjugated and unconjugated) | From Day 1 up to approximately 3 years
  This refers to the total amount of antibody present in a sample, regardless of whether it's attached to a drug (conjugated) or not (unconjugated). It includes a) Antibodies that are linked to the drug(conjugated antibodies) b) Antibodies that are not linked to any drug (unconjugated antibodies). This measurement gives an overall picture of the antibody concentration, which is important for understanding the pharmacokinetics of the ADC.
Module 1 and 2: Parts A and B: Plasma concentration of total unconjugated payload | From baseline up to approximately 3 years
  The "payload" typically refers to the cytotoxic drug that is attached to the antibody in an antibody drug conjugate (ADC).
  "Unconjugated payload" means the drug molecules that are not attached to any antibody.
  "Total unconjugated payload" refers to the total amount of free drug present in the sample.
  This measurement is crucial for assessing the stability of the ADC and understanding how much of the drug has been released from the antibody.
Module 1 and 2: Parts A and B: Change from baseline in STEAP2 tumour expression | From baseline up to approximately 3 years
  Target expression of STEAP2 will be evaluated using an analytically validated IHC assay.
Module 1 and 2: Parts A and B: Association of STEAP2 expression with AZD0516 response | From baseline up to approximately 3 years
  Expression of STEAP2 will be evaluated using an analytically validated IHC assay.
Module 1 and 2: Parts A and B: Number of participants with positive antidrug antibodies (ADAs) | Up to approximately 3 years
  To determine the immunogenicity of AZD0516 as monotherapy and in combination with anti-cancer agents.
Module 1: Part C: Number of participants with AEs, SAEs and AESIs | From Day 1 up to approximately 3 years
  To further assess the safety and tolerability of AZD0516 as monotherapy and in combination with anti-cancer agents.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (10):
  - Research Site, Fayetteville, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Providence, Rhode Island
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Houston, Texas
- Brazil (3):
  - Research Site, Barretos
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- China (3):
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Wuhan
- France (5):
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Saint-Herblain
  - Research Site, Suresnes
  - Research Site, Villejuif
- Italy (4):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kōtoku
- Poland (3):
  - Research Site, Koszalin
  - Research Site, Piotrkow Trybunalski
  - Research Site, Przemyśl
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Valencia
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Plymouth
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/